CLINICAL TRIAL: NCT06688760
Title: Endoscopic Nasopharyngectomy Combined with Retropharyngeal Lymph Node Dissection Plus Low-dose Radiotherapy Versus Bilateral Upper Neck Dissection for Newly Diagnosed Stage I Nasopharyngeal Carcinoma: a Randomized Controlled Clinical Trial
Brief Title: Surgery Alone Verus Sugery Combined with Dose-reduced Radiotherapy for Newly Diagnosed Stage I Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ming-Yuan Chen (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-sen University (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Huazhong University of Science and Technology Union Hospital (Nanshan Hospital) (Unknown); Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); First People's Hospital of Foshan (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Sponsor-Investigator, Ming-Yuan Chen, Professior,Chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2024-02-25
Record Dates: First submitted 2024-07-25; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-07

CONDITIONS: Nasopharyngeal Carcinoma; Surgery; Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery plus low dose radiotherapy (Experimental): Surgery:
  Endoscopic Nasopharyngectomy: Radical resection of primary lesion using nasal endoscopy.
  Retropharyngeal Lymphadenectomy: Radical retropharyngeal LNs resection using nasal endoscopy.
  Radiotherapy:
  Low Dose Raiotherapy:
  Low dose radiotherapy target area: CTV1: tumor bed area; For cases where the margin of the primary lesion is negative but less than 3mm, the margin area should be included; It should also include all cervical lymph nodes located above the cricoid cartilage detected by CT/MRI, regardless of size; CTV2: Low risk infiltration area.
  Intensity modulated radiation therapy prescription dose: CTV1: 36.00Gy/15Fr/2.40Gy; CTV2: 30.00Gy/15Fr/2.00Gy.
  Interventions: Procedure: Endoscopic nasopharyngectomy combine Retropharyngeal lymphadenectomy and Low Dose Radiotherapy
- Surgery (Experimental): Endoscopic Nasopharyngectomy: Radical resection of primary lesion using nasal endoscopy.
  Retropharyngeal Lymphadenectomy: Radical retropharyngeal LNs resection using nasal endoscopy.
  Bilateral Upper Neck Lymph Node Dissection: the specific cleaning area is the lymph nodes upon the Hyoid bone regions.
  Interventions: Procedure: Endoscopic nasopharyngectomy combine Retropharyngeal lymphadenectomy and Low Dose Radiotherapy; Procedure: Endoscopic nasopharyngectomy combine Retropharyngeal lymphadenectomy and Double upper neck lymph node dissection

INTERVENTIONS:
Procedure: Endoscopic nasopharyngectomy combine Retropharyngeal lymphadenectomy and Low Dose Radiotherapy — in experimental arm 1
Procedure: Endoscopic nasopharyngectomy combine Retropharyngeal lymphadenectomy and Double upper neck lymph node dissection — in experimental arm 2
  Arms: Surgery

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of endoscopic nasopharyngectomy combined with retropharyngeal lymph nodes dissection plus bilateral upper neck lymph node dissection or plus postoperative low-dose radiotherapy in newly diagnosed stage Ⅰ nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
At present, the newly diagnosed non metastatic nasopharyngeal carcinoma has achieved good therapeutic effect under the treatment scheme of intensity modulated radiotherapy. The 5-year survival rate of the newly diagnosed stage Ⅰ nasopharyngeal carcinoma was more than 95%. But at the same time, all patients receiving radical radiotherapy will experience different degrees of acute or chronic radiation injury, which will affect the quality of life of patients to varying degrees. For stage Ⅰ nasopharyngeal carcinoma with the primary lesion confined to the nasopharyngeal mucosa and without regional lymph node metastasis, in theory, the primary lesion can be removed by minimally invasive surgery without preventive treatment of cervical lymph nodes.

Our previous research results showed that endoscopic surgery could achieved similar survival outcomes but less adverse events than radiotherapy for Stage Ⅰ nasopharyngeal carcinoma with short diameter of retropharyngeal lymph nodes<0.4cm or short diameter of cervical lymph nodes<0.6 and negative PET/CT findings. However, if there is the same results for all stage I NPC patients is still unclear. Therefore, this study aims to compare the efficacy and safety of endoscopic nasopharyngectomy combined with retropharyngeal lymph node dissection combined with low-dose radiotherapy or bilateral upper neck lymph node dissection compared with conventional intensity-modulated radiotherapy.

When the patients participated in this study, the stage ⅠNPC patient of experimental group 1 received endoscopic nasopharyngectomy combined with retropharyngeal lymph node dissection and low-dose radiotherapy. Low dose radiotherapy target area: CTV1 (tumor bed area); For the primary lesion with negative margin but less than 3mm, the margin area should be included; For patients with extracapsular invasion of lymph nodes, the extracapsular invasion area should be included; It should also include all cervical lymph nodes located above the cricoid cartilage detected by CT/MRI, regardless of size; CTV2: low risk infiltration area. The prescription dose of intensity modulated radiotherapy: CTV1:36.00gy/15fr/2.40gy; CTV2:30.00gy/15fr/2.00gy. The patients in the stage Ⅰ in the experimental group 2 underwent endoscopic nasopharynx resection combined with retropharyngeal lymph node resection and bilateral upper neck lymph node dissection, without radiotherapy or chemotherapy after surgery.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Performance Status Score 0-1 points.
* Non-keratinized carcinoma of the nasopharynx (differentiated or undifferentiated, i.e., WHO type II or III) confirmed histologically and/or cytologically.
* According to the UICC/AJCC eighth edition staging, the patient is defined as T1N0M0 stage I.
* Adequate organ function: WBC ≥ 4×10^9 /L, NEUT ≥ 2×10^6 /L, HGB ≥ 9 g/dL, PLT count ≥ 100×10^9/L, TBIL ≤1.5 ULN, ALT ≤3 ULN, AST ≤3 ULN, ALP ≤3 ULN, ALB ≥ 3 g/dL, INR or APTT≤1.5 ULN, Scr ≤1.5 ULN or Ccr ≥ 60 mL/min.
* Informed Concent signed with willingness to obey the follow-up, treatment, examination and any other programs according to the research protocol.

Exclusion Criteria:

* Diagnosed as recurrent or distant metastatic nasopharyngeal carcinoma or together with any other malignancy.
* Suffering severe organ dysfunction or physical disorder which could not tolerate surgery or radiotherapy.
* Unable to cooperate with regular follow-up due to psychological, social, domestic or geological reasons.
* During pregnancy or lactation.
* Other patients that the chief physician considered as illegal for this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Local Regional Relapse-Free Survival (LRRFS) | 2 years
  The LRRFS is evaluated and calculated from the date of random assignment until the day of first local regional relapse or until the date of the last follow-up visit.

SECONDARY OUTCOMES:
The incidence of serious complications | 2 years
  Common Adverse Event Evaluation Criteria (CTCAE) version 5.0 evaluates acute and late-stage subjective toxicity reactions.
Overall Survival (OS) | 2 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Distant Metastasis-Free Survival (DMFS) | 2 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Progression-Free Survival (PFS) | 2 years
  The PFS was defined as the duration from the date of random assignment to the date of disease progression or censored at the date of the last follow-up.
Score of QLQ-C30 | 2 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ-C30) before treatment, during treatment, after treatment and follow up.
Score of H&N 35 | 2 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ-C30 and H&N 35) before treatment, during treatment, after treatment and follow up.
Incidence of acute postoperative complications | 2 weeks
  The incidence of acute postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — SUN yet-sen University
Locations (2):
- China (2):
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided